CLINICAL TRIAL: NCT02859935
Title: A SYNdemic BASed Co-located Linkage to Care INtervention for Men Who Have Sex With Men With High Risk Behavior: Design of a Randomized Controlled Trial
Brief Title: A SYNdemic BASed INtervention for MSM With High Risk Behavior: Design of a Randomized Controlled Trial
Acronym: SYNBASIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Public Health Service of Amsterdam (Other Government)
Responsible Party: Principal Investigator, Henry J.C. de Vries, Professor MD, PhD, Public Health Service of Amsterdam
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: synbasin 2.7
Record Dates: First submitted 2016-08-04; First posted 2016-08-09 (Estimated); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Risk Behavior
Keywords: HIV; drug abuse; MSM; Risk behavior; Sexually transmitted diseases; Sexually transmitted infections
MeSH Terms: conditions — Risk-Taking; Substance-Related Disorders; Sexually Transmitted Diseases | interventions — Mass Screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): The control group will receive standard care - 3 monthly STI screening, motivational interviewing and counselling. Both groups will get questionnaires on mental health problems: ADHD, depression, anxiety disorder, alexithymia and sex and drug addiction.
- Intervention group (Other): The intervention group will receive -besides standard care- additional questionnaires depending on their baseline questionnaires and in case of an indication for mental health problems, feedback and referral to relevant mental health and addiction care will be provided.
  Interventions: Behavioral: Screening and feedback

INTERVENTIONS:
Behavioral: Screening and feedback — Screening via questionnaires on mental health problems and feedback on the questionnaires
  Arms: Intervention group

SUMMARY:
The purpose of this randomized controlled intervention study at the STI outpatient clinic of Amsterdam is to answer the following questions : Does a personalised behaviour intervention comprising of targeted in-depth screening on mental health problems and drug use and, in case identified, subsequent linkage to care increase help seeking behaviour, and decrease risk behaviour in MSM who are at high risk for STIs and HIV?

ELIGIBILITY:
Inclusion Criteria:

* MSM
* Sufficient understanding of Dutch or English and
* 2 STIs in the last 24 months or a PEP treatment for HIV negative MSM

Exclusion Criteria:

* Men will be excluded if they are not able to complete follow-up or otherwise deemed by clinic staff to be unsuited for participation.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-09-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Help seeking behavior | one year
  Does a personalised behaviour intervention comprising of targeted in depth screening on mental health problems and drug use and linkage to care increase help seeking behaviour among MSM who are at high risk for STIs and HIV.

SECONDARY OUTCOMES:
Risk behavior | one year
  Does a behaviour intervention comprising of targeted in depth screening on mental health problems and drug use and linkage to care decrease STI prevalence and risky sex (i.e. condom use/ number of partners/ number of unsafe partners/ amount anal sex/ recreational drug use/ stop visiting the STI clinic).

CONTACTS AND LOCATIONS:
Overall Officials: Henry de Vries, MD, PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- STI Clinic, Public Health Service Amsterdam, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Achterbergh RCA, van Rooijen MS, van den Brink W, Boyd A, de Vries HJC. Enhancing help-seeking behaviour among men who have sex with men at risk for sexually transmitted infections: the syn.bas.in randomised controlled trial. Sex Transm Infect. 2021 Feb;97(1):11-17. doi: 10.1136/sextrans-2020-054438. Epub 2020 Jul 31. PMID 32737210
- [Derived] Achterbergh RCA, van der Helm JJ, van den Brink W, de Vries HJC. Design of a syndemic based intervention to facilitate care for men who have sex with men with high risk behaviour: the syn.bas.in randomized controlled trial. BMC Infect Dis. 2017 Jun 6;17(1):398. doi: 10.1186/s12879-017-2474-x. PMID 28587607